CLINICAL TRIAL: NCT05597891
Title: A Safety and Feasibility Single-Arm Study of a Novel Catheter Thrombectomy Device For the Treatment of Pulmonary Embolism (ENGULF)
Brief Title: Endovascular Engineering ENGULF Study
Acronym: ENGULF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endovascular Engineering (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN01001
Record Dates: First submitted 2022-10-14; First posted 2022-10-28 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational Device (Experimental): The study design includes two cohorts: a Pre-Pivotal Cohort of up to 50 subjects (25 Feasibility and up to 25 Roll-Ins), and a Pivotal Cohort enrolling up to 131 subjects, to yield 100 evaluable subjects at 48 hours post procedure.
  Interventions: Device: Hēlo PE Thombectomy System

INTERVENTIONS:
Device: Hēlo PE Thombectomy System — Treatment with the Hēlo PE Thombectomy System for thromboembolectomy

SUMMARY:
Evaluation of initial safety and clinical feasibility of the Hēlo PE Thrombectomy System for thrombectomy in acute submassive pulmonary embolism (PE).

ELIGIBILITY:
Asterisks * indicate entry criteria that can be evaluated during prescreening without obtaining informed consent as they are part of standard of care PE management. Asterisks in parenthesis (*) indicate entry criteria that can be evaluated during prescreening without obtaining informed consent at Sites that routinely perform CTA as part of standard of care in PE management.

Inclusion Criteria:

Patients must meet ALL of the following criteria to be eligible for participation in the study:

1. *Patient is > 18 and < 90 years old
2. *Clinical signs and symptoms consistent with acute submassive PE with duration ≤ 14 days, as determined by the Investigator
3. (*)CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery)
4. (*)RV/LV ratio of ≥ 0.9 (Enrollment qualification assessment based on Investigator's interpretation of RV/LV ratio at baseline)
5. *Systolic blood pressure ≥ 90 mmHg (initial SBP may be ≥ 80 mmHg if the pressure recovers to ≥ 90 mmHg with fluids)
6. *Heart rate < 130 BPM prior to procedure
7. *Patient is deemed medically eligible for interventional procedure(s), per investigator guidelines and clinical judgment
8. Patient signs a written Informed Consent form to participate in the study, prior to any study mandated procedures

Exclusion Criteria:

Patients must be EXCLUDED from participation in this study if ANY of the following criteria are met:

1. *Acute massive PE at presentation
2. *Prior PE within last 6 months
3. *Thrombolytic use within 30 days of baseline CTA
4. *Pulmonary hypertension with peak pulmonary artery systolic pressure > 70 mmHg by right heart catheterization
5. *Vasopressor requirement after fluids to keep pressure ≥ 90 mmHg
6. *FiO2 requirement > 40% or > 6 LPM to keep oxygen saturation > 90%
7. *Hematocrit < 28% (NOTE: hematocrit required within 24 hours of index procedure)
8. *Platelets < 100,000/μL
9. *Serum creatinine > 1.8 mg/dL
10. *International normalized ratio (INR) > 3
11. *aPTT (or PTT) > 50 seconds on no anticoagulation
12. *Major trauma < 14 days
13. *Presence of intracardiac lead in the right ventricle or right atrium placed within 6 months
14. *Cardiovascular or pulmonary surgery within last 7 days
15. *Life expectancy less than 1 year due to advanced malignancy, as determined by the investigator at the time of enrollment
16. *Known bleeding diathesis or coagulation disorder
17. *Known left bundle branch block
18. *History of severe pulmonary arterial hypertension
19. *History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
20. *History of uncompensated heart failure
21. *History of underlying lung disease that is oxygen dependent
22. *Presence of IVC filter and or iliocaval stents
23. *History of heparin-induced thrombocytopenia (HIT)
24. *Any contraindication to systemic or therapeutic doses of heparin or anticoagulants
25. *Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
26. *Known allergy to any device component
27. (*)Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the Subject is not appropriate for mechanical thrombectomy intervention (e.g., inability to navigate to target location, predominately chronic clot or non-clot embolus)
28. *Life expectancy of < 90 days, as determined by Investigator
29. *Female who is pregnant or nursing
30. *Current participation in another investigational drug or device treatment study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Objective | 48 hours following the procedure
  Composite device-related Major Adverse Event (MAE) rate, defined as any of the following events within 48 hours (+/- 24 hours) of the procedure:
  * Death
  * Life-threatening, disabling or major bleeding as defined by VARC-2
  * Serious adverse events, including, clinical deterioration, pulmonary vascular injury, and cardiac injury
Primary Performance Objective | 48 hours following the procedure
  Clinical Success, defined as the reduction in RV/LV ratio from baseline to 48 hours (+/- 24 hours, or discharge, whichever occurs first) as assessed by CTA

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Klein, MD, Principal Investigator — Piedmont Heart; Julie Bulman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (19):
- United States (19):
  - Huntington Hospital, Pasadena, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Delray Medical Center, Delray Beach, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - HCA Florida Memorial Hospital, Jacksonville, Florida
  - Piedmont Heart, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - TriHealth Hatton Research Institute, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Wellmont Cardiology Services / Ballad Health, Kingsport, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Austin Heart, Austin, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - UT Health, Houston, Texas
  - Gundersen Health, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No